CLINICAL TRIAL: NCT03039582
Title: Short Anovaginal Distance is Associated With Obstetric Anal Sphincter Rupture
Acronym: AVD and OASR
Status: Completed | Type: Observational
Sponsor: Ostergotland County Council, Sweden (Other)
Responsible Party: Principal Investigator, Eva Uustal, Senior consultant, Ostergotland County Council, Sweden
Other Study IDs: OstergotlandCC2
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Perineal Tear; Obstetric Trauma
Keywords: perineal tear; bidigital palpation; perineal ultrasound; post partum diagnostics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Probable grad 2: Perineal laceration Probable grad 2
  Interventions: Diagnostic Test: Bidigital palpation; Diagnostic Test: Perineal ultrasound
- Suspected grade 3: Perineal laceration Suspected grade 3
  Interventions: Diagnostic Test: Bidigital palpation; Diagnostic Test: Perineal ultrasound
- Probable grad 3: Perineal laceration Probable grad 3
  Interventions: Diagnostic Test: Bidigital palpation; Diagnostic Test: Perineal ultrasound

INTERVENTIONS:
Diagnostic Test: Bidigital palpation — palpation of the anovaginal distance with two fingers
Diagnostic Test: Perineal ultrasound — ultrasound measurement of the anovaginal distance
  Other Names: Vaginal ultrasound; transperineal ultrasound

SUMMARY:
Anovaginal distance measured by palpation and perineal ultrasound are similar.

DETAILED DESCRIPTION:
Background: Objective diagnostic methods for obstetric anal sphincter rupture, (OASR) such as endoanalt ultrasound (EAUS), show missed ruptures that can lead to anal incontinence. To perform EAUS after all deliveries at all hours, although it may lead to diagnostic improvement is not feasible in most delivery wards. Another objective method for screening women after delivery to identify OASR would be of value. Bidigital palpation of the perineum is often suggested without specifying what results are relevant.

AIM:

The aim of this study was to establish if the palpated anovaginal distance after delivery could be confirmed by perineal ultrasound and correlated to the extent of the perineal tear.

MATERIALS AND METHODS:

A structured educational programme for midwives (palpation) and doctors (perineal ultrasound) was accomplished. Midwives were instructed to record the palpated anovaginal distance in primiparae with spontaneous vaginal delivery and no episiotomy. If the AVD was found to be shorter than 2 cm, she recorded a primary diagnosis of probable grade 2, suspected grade 3 or probable grade 3 and called the doctor. The AVD was then measured by perineal ultrasound by a doctor aware of a laceration but not it´s extent, which was then established by clinical exam and perineal ultrasound.

ELIGIBILITY:
Inclusion Criteria: women who just had their firstborn child through vaginal delivery at the delivery ward at the University Hospital in Linköping, Sweden from October 2014 to January 2016.

-

Exclusion Criteria: inability to understand swedish

-

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women just after vaginal delivery
Sampling Method: Non-Probability Sample
Enrollment: 151 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2016-01-31 (Actual); Study Completion 2017-01-19 (Actual)

PRIMARY OUTCOMES:
Correlation between palpated and ultrasound- measured anovaginal distance | immediate
  Does palpation give a reliable result?

SECONDARY OUTCOMES:
Anal Sphincter rupture incidence | immediate
  How common is anal sphincter rupture

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harvey MA, Pierce M, Alter JE, Chou Q, Diamond P, Epp A, Geoffrion R, Harvey MA, Larochelle A, Maslow K, Neustaedter G, Pascali D, Pierce M, Schulz J, Wilkie D, Sultan A, Thakar R; Society of Obstetricians and Gynaecologists of Canada. Obstetrical Anal Sphincter Injuries (OASIS): Prevention, Recognition, and Repair. J Obstet Gynaecol Can. 2015 Dec;37(12):1131-48. doi: 10.1016/s1701-2163(16)30081-0. PMID 26637088
- [Background] Geller EJ, Robinson BL, Matthews CA, Celauro KP, Dunivan GC, Crane AK, Ivins AR, Woodham PC, Fielding JR. Perineal body length as a risk factor for ultrasound-diagnosed anal sphincter tear at first delivery. Int Urogynecol J. 2014 May;25(5):631-6. doi: 10.1007/s00192-013-2273-x. Epub 2013 Dec 12. PMID 24337585
- [Background] Santoro GA, Wieczorek AP, Dietz HP, Mellgren A, Sultan AH, Shobeiri SA, Stankiewicz A, Bartram C. State of the art: an integrated approach to pelvic floor ultrasonography. Ultrasound Obstet Gynecol. 2011 Apr;37(4):381-96. doi: 10.1002/uog.8816. PMID 20814874
- [Background] Shobeiri SA, Nolan TE, Yordan-Jovet R, Echols KT, Chesson RR. Digital examination compared to trans-perineal ultrasound for the evaluation of anal sphincter repair. Int J Gynaecol Obstet. 2002 Jul;78(1):31-6. doi: 10.1016/s0020-7292(02)00068-1. PMID 12113968